CLINICAL TRIAL: NCT00005864
Title: A Phase II Study of Chloroquinoxaline Sulfonamide (CQS) in Colorectal Cancer Stage IV
Brief Title: Chloroquinoxaline Sulfonamide in Treating Patients With Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067896; OSU-NCI-56; NCI-56
Record Dates: First submitted 2000-06-02; First posted 2004-02-25 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2002-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — 5-chloroquinoxaline-2-sulfanilamide

INTERVENTIONS:
Drug: chloroquinoxaline sulfonamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of chloroquinoxaline sulfonamide in treating patients who have stage IV colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity and toxicities of chloroquinoxaline sulfonamide in patients with stage IV colorectal cancer.

OUTLINE: This is a multicenter study. Patients receive chloroquinoxaline sulfonamide IV over 1 hour weekly for 4 consecutive weeks. Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed for at least 30 days.

PROJECTED ACCRUAL: A total of 16-25 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IV colorectal cancer Measurable disease defined as lesions that measure at least 20 mm in one dimension using conventional techniques or at least 10 mm with spiral CT scan not including: Bone lesions Leptomeningeal disease Ascites Pleural/pericardial effusion Inflammatory breast disease Lymphangitis cutis/pulmonis Abdominal masses that are not confirmed and followed by imaging techniques Cystic lesions Recurrent disease allowed after adjuvant chemotherapy if recurrence occurred at least 6 months after completion of therapy No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 60-100% Life expectancy: Greater than 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST/ALT no greater than 2.5 times upper limit of normal Renal: Creatinine normal Cardiovascular: No history of symptomatic congestive heart failure, unstable angina, or cardiac arrhythmia (e.g., supraventricular tachycardia or atrial fibrillation) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No significant episodes of hypoglycemia in past 6 months No known allergies to compounds of similar chemical or biologic composition to chloroquinoxaline sulfonamide No known glucose-6 phosphate deficiency or hemolytic anemia No uncontrolled concurrent illness (e.g., active infection) No concurrent psychiatric illness or social condition that would preclude compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: One prior biologic therapy allowed Chemotherapy: See Disease Characteristics No more than one prior chemotherapy for metastatic disease or adjuvant treatment At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered Endocrine therapy: No concurrent oral hypoglycemics or insulin Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified Other: No other concurrent investigational agents No concurrent combination antiretroviral treatment for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric H. Kraut, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio